CLINICAL TRIAL: NCT00042549
Title: Biliary Lithotripsy in Combination With Actigall Versus Actigall Monotherapy for the Treatment of Symptomatic Cholesterol Gallstones
Brief Title: Lithotripsy for the Treatment of Gallstones
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Medstone International (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GS-PA-001
Record Dates: First submitted 2002-07-31; First posted 2002-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Cholelithiasis
Keywords: Gallstones; Gallstone; Biliary stones; Gallbladder stones; Gallbladder; Lithotripsy; Cholelithiasis; ESWL; Shock wave; Shock waves; shockwaves; shockwave
MeSH Terms: conditions — Cholelithiasis; Gallstones; Cholecystolithiasis | interventions — Lithotripsy; Ursodeoxycholic Acid

INTERVENTIONS:
Device: Extracorporeal Shock Wave Lithotripsy
Drug: ursodiol

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of using the Medstone lithotripter to treat single non-calcified gallstones from 4 to 20 mm in diameter.

DETAILED DESCRIPTION:
This study is a randomized, single-masked controlled trial in which the combination therapy of lithotripsy and the bile acid drug Actigall is compared to monotherapy with only Actigall. The primary objectives are, 1) To determine whether the use of the Medstone STS Lithotripter system in combination with the orally administered drug Actigall is more effective (as measured by percentages of stone free patients 6 months after randomization) in reducing single non-calcified radiolucent gallstones (from 4 to 20mm in diameter) than use of Actigall alone, and 2) To demonstrate that use of the Medstone lithotripsy system is safe (as measured by incidence of adverse events) for the intended purpose, when operated according to its labeling.

ELIGIBILITY:
* History of biliary pain
* Evidence of a single noncalcified, radiolucent gallstone between 4 and 20 mm (inclusive) diameter
* HIDA scan demonstrating patency of cystic bile duct
* No cardiac pacemaker
* No allergy to radioopaque dye, iodine, bile acids
* No spontaneous or iatrogenic bleeding disorder
* No current or prior bile duct obstruction, cholangitis, pancreatitis, or cholecystitis
* Not pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Ertan, M.D., Study Director — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - The Methodist Hospital, Houston, Texas
  - Virgina Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Ertan A. Treatment of gallstones by extracorporeal shock wave lithotripsy. Am J Gastroenterol. 2002 Apr;97(4):831-2. doi: 10.1111/j.1572-0241.2002.05738.x. No abstract available. PMID 12003415
- [Background] Ertan A, Hernandez RE, Campeau RJ, Geshner JR, Litwin MS. Extracorporeal shock-wave lithotripsy and ursodiol versus ursodiol alone in the treatment of gallstones. Gastroenterology. 1992 Jul;103(1):311-6. doi: 10.1016/0016-5085(92)91128-q. PMID 1612339
- [Background] Vanderpool D, Jones RC, O'Leary JP, Hamilton JK. Biliary lithotripsy. Am J Surg. 1989 Sep;158(3):194-7. doi: 10.1016/0002-9610(89)90251-1. PMID 2672841
- [Background] Sackmann M, Pauletzki J, Sauerbruch T, Holl J, Schelling G, Paumgartner G. The Munich Gallbladder Lithotripsy Study. Results of the first 5 years with 711 patients. Ann Intern Med. 1991 Feb 15;114(4):290-6. doi: 10.7326/0003-4819-114-4-290. PMID 1987875
- [Background] Pelletier G, Raymond JM, Capdeville R, Mosnier H, Caroli-Bosc FX. Gallstone recurrence after successful lithotripsy. J Hepatol. 1995 Oct;23(4):420-3. doi: 10.1016/0168-8278(95)80200-2. PMID 8655959
- See also: UpToDate is a practical clinical information service (always current). It is written by a recognized faculty of experts who each address a specific clinical issue. They synthesize the latest evidence and best practices. — http://patients.uptodate.com/frames.asp?page=tocmain.asp